CLINICAL TRIAL: NCT03044522
Title: A Multicenter Study Comparing the Patient Outcomes Associated With Use of a Nurse Pain Educator for Patients With Chronic Pain
Brief Title: Use of a Nurse Pain Educator for Patients With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NEMA Research, Inc. (Industry)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NEMA-SUPeR-001
Record Dates: First submitted 2017-02-01; First posted 2017-02-07 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Chronic Pain; Opioid Use; Nurse's Role
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Nurse Education (No Intervention): Subjects who are enrolled into study arm with no Nurse Pain Educator will be monitored every month to assess their use of their medication, quality of life, physical and mental well-being. No intervention will be conducted with these subjects beyond that of standard of care at the facility.
- Nurse Education (Other): Subject enrolled into the Nurse Pain Educator arm will be educated (Opioid Education) on different opioid pain management topics with a focus on safe and appropriate use and consumption of opioid analgesics.
  Interventions: Other: Opioid Education

INTERVENTIONS:
Other: Opioid Education
  Arms: Nurse Education

SUMMARY:
This multicenter randomized (block randomization) controlled parallel arm pilot study comparing the incorporation vs no incorporation of a Nurse Pain Educator into clinics that treat chronic non cancer pain patients with opioid analgesics. Subjects who are either opioid naïve or opioid experienced will be enrolled into the study.

DETAILED DESCRIPTION:
The Nurse Pain Educator arm shall have two phases: a Pre-Teaching Phase and a Teaching/Knowledge Maintenance Phase. During the Pre-Teaching Phase, all subjects who are enrolled will complete different baseline assessments and will be prescribed an opioid. Subjects will then enter the Teaching/Knowledge Maintenance Phase. Subject enrolled into the Nurse Pain Educator arm will be educated on different opioid pain management topics with a focus on safe and appropriate use and consumption of opioid analgesics. Subjects will meet monthly with the Nurse Educator for up to 5 months for reinforcement of their training and to assess their use of their medication, their quality of life and their physical and mental well-being.

Subjects who are enrolled into the study arm with no Nurse Pain Educator will be monitored every month to assess their use of their medication, their quality of life and their physical and mental well-being. No intervention will be conducted with these subjects beyond that of standard of care at the facility. Subjects will be evaluated monthly but primary differences in outcomes will compare baseline to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read, understand, and provide written informed consent
* Male or Female patients ≥ 18 years of age
* Diagnosed with non-cancer pain for >3 months
* Ability to meet study requirements (i.e., can attend monthly visits, able to complete questionnaires, etc.)
* Prescribed an oral opioid that will last duration of the study period
* Provide a completed Opioid Patient Prescriber Agreement

Exclusion Criteria:

* Diagnosed with chronic cancer pain
* Personal or family history of alcohol or drug abuse in the past 5 years
* Personal or family history of major mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2017-09-21 (Actual); Study Completion 2017-11-21 (Actual)

PRIMARY OUTCOMES:
Change in Opioid Consumption | 6 Months
  Difference between opioid consumption in subjects with and without education by a Nurse Pain Educator as measured by Total Morphine Sulfate Equivalent of Prescription from change in baseline to end of study and at each month.
Change Opioid Consumption | 6 Months
  Difference between opioid consumption in subjects with and without education by a Nurse Pain Educator as measured by a Qualitative Assessment of Opioid consumption from change in baseline to end of study and at each month.

SECONDARY OUTCOMES:
Change in Current Opioid Misuse Measure (COMM) | 6 Months
  Assess Safe and Appropriate Use of Opioids by measuring change in Currenet Opioid Misuse Measure from baseline to end of study and at each month.
Change in Pain Medicine Questionnaire (PMQ) | 6 Months
  Assess Safe and Appropriate Use of Opioids by measuring change in Pain Medicine Questionnaire from baseline to end of study and at each month.
Change in SF-36 | 6 Months
  Assess Quality of Life and Daily Function by measuring the change in the SF-36 Health Outcomes survey from baseline to end of study and at each month.
Change in Quality of Life Scale | 6 Months
  Assess Quality of Life and Daily Function by measuring the change in the 11 point Quality of Life Scale from baseline to end of study and at each month.

OTHER OUTCOMES:
Online Pain Assessment Tool | 6 Months
  Assess ease of use and outcomes of the Online Pain Assessment Tool from change in baseline to end of study in the Online Pain Assessment Tool scores

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Pergolizzi, MD, Principal Investigator — NEMA Research, Inc.
Locations (4):
- United States (4):
  - Headache and Pain Management Center of SWFL, Fort Myers, Florida
  - Gold Coast Research, Plantation, Florida
  - Mid America Physiatrists, Overland Park, Kansas
  - Piedmont Family Practice, Warrenton, Virginia

IPD SHARING:
Plan to Share IPD: No
The data will be presented in a manuscript/publication in a peer-reviewed journal.